CLINICAL TRIAL: NCT06302374
Title: A Multicentre, Randomized, Double-Blind, Placebo-Controlled, Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of GR2001 Injection in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of GR2001 in Chinese Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GR2001-001
Record Dates: First submitted 2024-02-28; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Tetanus
MeSH Terms: conditions — Tetanus | interventions — Tetanus Toxoid

STUDY DESIGN:
Intervention Model Description: In the phase I part of the study, a total of 94 healthy subjects will be enrolled. The 94 healthy adult subjects will be enrolled into 7 cohorts sequentially. Each participant will receive a single IM dose of GR2001 or placebo or HTIG according to the cohort in which they were enrolled. After injection (Day 0), participants will remain in the study site for observation up to Day 1. The phase I part will last for 105 days following the assessments of safety, PK, PD and ADA.
  In the phase II part of the study, a total of 108 healthy subjects will be enrolled. The 108 healthy subjects will be randomly assigned to the experimental group and the control group based on a ratio of 1:1:1:2:2:2.The phase II part will last for 105 days following the assessments of safety, PK, PD and ADA.
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort 1 GR2001 0.01mg/kg/placebo (Experimental): Four subjects will be randomly assigned to receive either GR2001 or placebo at a 3:1 ratio (i.e. 3 subjects receive GR2001 and 1 with placebo).
  Interventions: Biological: GR2001; Biological: Placebo
- Cohort 2 GR2001 0.02mg/kg/placebo (Experimental): Ten subjects will be randomly assigned to receive either GR2001 or placebo at a 4:1 ratio (i.e. 8 subjects receive GR2001 and 2 with placebo).
  Interventions: Biological: GR2001; Biological: Placebo
- Cohort 3 GR2001 0.05mg/kg/placebo/HTIG (Experimental): 24 subjects will be randomly assigned to receive GR2001 or placebo or HTIG(250IU) at a 1:1:1 ratio (i.e. 8 subjects receive GR2001, 8 with placebo and 8 with HTIG).
  Interventions: Biological: GR2001; Biological: Placebo; Biological: HTIG
- Cohort 4 GR2001 0.1mg/kg/placebo (Experimental): Ten subjects will be randomly assigned to receive either GR2001 or placebo at a 4:1 ratio (i.e. 8 subjects receive GR2001 and 2 with placebo).
  Interventions: Biological: GR2001; Biological: Placebo
- Cohort 5 GR2001 0.2mg/kg/placebo (Experimental): Ten subjects will be randomly assigned to receive either GR2001 or placebo at a 4:1 ratio (i.e. 8 subjects receive GR2001 and 2 with placebo).
  Interventions: Biological: GR2001; Biological: Placebo
- Cohort 6 GR2001 0.1mg/kg/placebo (Experimental): Eighteen subjects will be randomly assigned to receive either GR2001 or placebo at a 2:1 ratio (i.e. 12 subjects receive GR2001 and 6 with placebo) followed by a dose of Tetanus Toxoid（TT） on Day0.
  Interventions: Biological: GR2001; Biological: Placebo; Biological: Tetanus Toxoid
- Cohort 7 GR2001 0.2mg/kg/placebo (Experimental): Eighteen subjects will be randomly assigned to receive either GR2001 or placebo at a 2:1 ratio (i.e. 12 subjects receive GR2001 and 6 with placebo) followed by a dose of Tetanus Toxoid（TT） on Day0.
  Interventions: Biological: GR2001; Biological: Placebo; Biological: Tetanus Toxoid
- Cohort 8 GR2001 0.1mg/kg/ GR2001 0.2mg/kg/ HTIG (Experimental): Thirty six subjects will be randomly assigned to receive GR2001(0.1mg/kg) or GR2001(0.2mg/kg) or HTIG(250IU) at a 1:1:1 ratio (i.e. 12 subjects receive GR2001(0.1mg/kg), 12 with GR2001(0.2mg/kg) and 12 with HTIG).
  Seventy two subjects will be randomly assigned to receive GR2001(0.1mg/kg) or GR2001(0.2mg/kg) or HTIG(250IU) at a 1:1:1 ratio (i.e. 24 subjects receive GR2001(0.1mg/kg), 24 with GR2001(0.2mg/kg) and 24 with HTIG) followed by one dose of Tetanus Toxoid（TT） on Day0 and Day28.
  Interventions: Biological: GR2001; Biological: HTIG; Biological: Tetanus Toxoid

INTERVENTIONS:
Biological: GR2001 — intramuscular injection
Biological: Placebo — intramuscular injection
  Arms: Cohort 1 GR2001 0.01mg/kg/placebo; Cohort 2 GR2001 0.02mg/kg/placebo; Cohort 3 GR2001 0.05mg/kg/placebo/HTIG; Cohort 4 GR2001 0.1mg/kg/placebo; Cohort 5 GR2001 0.2mg/kg/placebo; Cohort 6 GR2001 0.1mg/kg/placebo; Cohort 7 GR2001 0.2mg/kg/placebo
Biological: HTIG — intramuscular injection
  Arms: Cohort 3 GR2001 0.05mg/kg/placebo/HTIG; Cohort 8 GR2001 0.1mg/kg/ GR2001 0.2mg/kg/ HTIG
Biological: Tetanus Toxoid — intramuscular injection
  Arms: Cohort 6 GR2001 0.1mg/kg/placebo; Cohort 7 GR2001 0.2mg/kg/placebo; Cohort 8 GR2001 0.1mg/kg/ GR2001 0.2mg/kg/ HTIG

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and Immunogenicity characteristics of GR2001 and compare the anti-tetanus neutralizing antibody titers of GR2001 with human tetanus immunoglobulin (HTIG)in healthy adult subjects.

DETAILED DESCRIPTION:
This is a Multicentre, Randomized, Double-Blind, Placebo-Controlled, Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of GR2001 Injection in Healthy Subjects.

In the phase I part of the study, a total of 94 healthy subjects will be enrolled. The 94 healthy adult subjects will be enrolled into 7 cohorts sequentially. Each participant will receive a single IM dose of GR2001 or placebo or HTIG according to the cohort in which they were enrolled. After injection (Day 0), participants will remain in the study site for observation up to Day 1. The phase I part will last for 105 days following the assessments of safety, PK, PD and ADA.

In the phase II part of the study, a total of 108 healthy subjects will be enrolled. The 108 healthy subjects will be randomly assigned to the experimental group and the control group based on a ratio of 1:1:1:2:2:2.The phase II part will last for 105 days following the assessments of safety, PK, PD and ADA.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, 18-60 years of age (both inclusive);
2. Body mass index within 18.0-27.0 kg/m2 (both inclusive);
3. Subjects including partners are willing to voluntarily take effective contraceptive measures from screening to 6 months after the last study drug administration.
4. Completed written informed consent process, signed the informed consent forms and Agreed to complete all follow-ups.

Exclusion Criteria:

1. History or evidence of severe drug or excipient allergy;
2. History or evidence of tetanus infection;
3. Inoculation of tetanus vaccine within 10 years;
4. History or evidence of any other acute or chronic disease；
5. Known or suspected history of drug abuse；
6. Positive outcome for Tetanus-antibody IgG test;
7. Nursing mothers or pregnant women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2023-03-04 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs(Phase I) | Up to 105 days
  Number of participants with treatment-related adverse events or serious adverse events.
Tetanus-antibody titer(Phase II) | 24 hours post administration
  Tetanus-antibody titer post administration.

SECONDARY OUTCOMES:
Tetanus-antibody titer(Phase I/II) | Up to 105 days
  Tetanus-antibody titer post administration.
Incidence of ADA(Phase I/II) | Up to 105 days
  Incidence of ADA post administration.
Incidence of AEs(Phase II) | Up to 105 days
  Number of participants with treatment-related adverse events or serious adverse events.
Peak plasma concentration(Cmax) | Up to 105 days
  Estimated by non-compartmental analysis (NCA) with WinNonlin.
Area under the plasma concentration versus time curve (AUC) | Up to 105 days
  Estimated by non-compartmental analysis (NCA) with WinNonlin.
Time of maximum plasma concentration (Tmax) | Up to 105 days
  Estimated by non-compartmental analysis (NCA) with WinNonlin.
Terminal half-life (T1/2) | Up to 105 days
  Estimated by non-compartmental analysis (NCA) with WinNonlin.
Apparent total body clearance (CL/F) | Up to 105 days
  Estimated by non-compartmental analysis (NCA) with WinNonlin.
Apparent volume of distribution (Vd/F) | Up to 105 days
  Estimated by non-compartmental analysis (NCA) with WinNonlin.
The elimination rate constant (Kel) | Up to 105 days
  Estimated by non-compartmental analysis (NCA) with WinNonlin.
Mean Residence Time (MRT) | Up to 105 days
  Estimated by non-compartmental analysis (NCA) with WinNonlin.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, PHD, Principal Investigator — Huashan Hospital affiliated of Fudan University
Locations (1):
- Huashan Hospital affiliated of Fudan University, Shanghai, Shanghai Municipality, China